CLINICAL TRIAL: NCT00089830
Title: A Safety and Efficacy Study of MSI-1256F (Squalamine Lactate) To Treat "Wet" Age-Related Macular Degeneration
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Genaera Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSI-1256F-209
Record Dates: First submitted 2004-08-16; First posted 2004-08-17 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Macular Degeneration
Keywords: Subfoveal Choroidal Neovascularization; Squalamine Lactate
MeSH Terms: conditions — Macular Degeneration | interventions — squalamine lactate

INTERVENTIONS:
Drug: MSI-1256F (Squalamine Lactate)

SUMMARY:
Age-Related Macular Degeneration (AMD) is a degenerative eye disease of the retina that causes a progressive loss of central vision. AMD is the leading cause of legal blindness among adults age 50 or older in the Western world. AMD presents in two different types - "dry" and the more severe "wet" form. Wet AMD is caused by the growth of abnormal blood vessels in the macula. Squalamine lactate is an investigational drug that may prevent the growth of these abnormal blood vessels. This study will test the safety and efficacy of Squalamine in the treatment of AMD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of "wet" age-related macular degeneration

Exclusion Criteria:

* Prior treatment of "wet" age-related macular degeneration in the affected eye in the past 3 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-08; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Genaera Corporation, Plymouth Meeting, Pennsylvania, United States